CLINICAL TRIAL: NCT07053943
Title: Revision Rate Due to Infection With Single-dose Versus Multiple-dose Antibiotic Prophylaxis During Primary Hip- and Knee Arthroplasty: A Hybrid Effectiveness Implementation Target Trial Emulation Study.
Brief Title: Infection-related Revision Rates After Single-dose Versus Multiple-dose Antibiotic Prophylaxis in Primary Hip and Knee Arthroplasty: a Comparative Implementation Study.
Acronym: REVISE
Status: Enrolling by invitation | Type: Observational
Sponsor: JointResearch (Other)
Collaborators: Dutch Arthroplasty Register (LROI) (Unknown)
Responsible Party: Sponsor
Other Study IDs: WO 25.069
Record Dates: First submitted 2025-06-23; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Total Hip Arthroplasty (THA); Antibiotic Prophylaxis; Revision Arthroplasty; Total Knee Arthroplasty
Keywords: Antibiotic Prophylaxis; Total Knee Arthroplasty; Total hip Arthroplasty; revision Arthroplasty

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Single-dose antibiotic prophylaxis in Total Hip Arthroplasty: All patients undergoing Total Hip Arthroplasty before the guideline advocating for a multiple dose antibiotic regime.
- Single-dose antibiotic prophylaxis in Total Knee Arthroplasty: All patients undergoing Total Knee Arthroplasty before the guideline advocating for a multiple dose antibiotic regime.
- Multi-dose antibiotic prophylaxis in Total Hip Arthroplasty: All patients undergoing Total Hip Arthroplasty after the guideline advocating for a multiple dose antibiotic regime.
- Multi-dose antibiotic prophylaxis in Total Knee Arthroplasty: All patients undergoing Total Hip Arthroplasty after the guideline advocating for a multiple dose antibiotic regime.

SUMMARY:
Prosthetic Joint Infection (PJI) is a significant issue in joint replacement surgeries, causing additional surgeries and substantial healthcare costs. An effective way of preventing these infections is through the use of antibiotics before and after surgery. However, there is ongoing debate regarding the optimal dosage regimen for these antibiotics to achieve maximum effectiveness. In the Netherlands, most hospitals currently give multiple doses of antibiotics for hip and knee replacement surgeries. A new upcoming guideline recommends using only one dose of antibiotics, which could have several benefits. It might reduce the need for antibiotics overall, decrease the work for nurses, and shorten hospital stays. However, it is unclear if this change is safe or effective.

This study aims to compare the effectiveness of the current multi-dose antibiotic method with the new single-dose approach. We will also look at how well hospitals adopt this new guideline (implementation) and compare the healthcare costs associated with both antibiotic regimens. By studying real-world data from surgeries and patient records, we want to determine if the single-dose strategy is as effective at preventing infections and reducing the need for additional surgeries.

DETAILED DESCRIPTION:
SUMMARY Rationale: Antibiotic Stewardship (AS) is focusing on the precise use of antibiotics to enhance patient outcomes and curb antibiotic resistance. This concept is especially pertinent in the context of Prosthetic Joint Infection (PJI), a primary cause for revision hip arthroplasty (RHA) and revision knee arthroplasty (RKA). While perioperative antibiotic prophylaxis has proven to significantly reduce PJI risk, the optimal duration-whether to administer a single dose or multiple doses-remains hotly debated. When reflecting on the administration practices, a 2018 national survey indicated that 90% of Dutch hospitals utilized multi-dose antibiotic prophylaxis during total hip arthroplasty (THA) and total knee arthroplasty (TKA). The Federation for Medical Specialisten (FMS) reviewed the perioperative antibiotic prophylaxis guideline to more strongly endorse single-dose prophylaxis. By evaluating implementation effectiveness following the updated guideline and assessing the broader implications on healthcare costs, this study seeks to deliver insights that could shape future antibiotic use in orthopaedic surgery, ultimately influencing policies and practices in the Netherlands and beyond.

Objective: The objectives of the study are as follows:

1. Assess the implementation-effectiveness of the single-dose implementation strategy following the new guideline's introduction by assessing the percentage of hospitals that adopt to the new guideline and the time these hospitals take to do so.
2. Compare the rate of revision procedures due to infection between single-dose and multiple-dose antibiotic prophylaxis during THA and TKA by comparing the relative amount of revisions surgeries due to infection one year before implementation of the new guideline and one year after implementation of the new guideline.
3. Compare the healthcare costs between single-dose and multi-dose perioperative antibiotic prophylaxis by estimating the cost per antibiotic dose and the costs related to the extended hospital admission.

Study design: A novel hybrid, non-inferiority, de-implementation effectiveness target trial emulation study using real-world data is proposed to complete the study objectives:

1. A survey will be sent to orthopaedic surgeons from Dutch institutions performing THA and TKA. The questions relate to their current antibiotic policy and their intention to adopt to the new guideline. Institutions that comply with the current guideline and intent to adopt the new guideline within the next year will be included. The included Institutions will be actively monitored to determine the successfulness of the implementation of the single-dose prophylaxis strategy.
2. Data from the Dutch arthroplasty register (LROI) will be used to document the relative amount of revision procedures due to infection for all included institutions. The relative amount of revision procedures for infection will be compared between the year before adoption to the new guideline and the year after.
3. Innovative search software (CTcue) will be employed to retrieve individual patient data from electronic patient records for all patients who underwent THA or TKA in the observation period. 4. 4. The data from the LROI register (institution level) will be compared to the data retrieved from electronic patient records by CTcue (patient level). In this way, we aim to validate the LROI database regarding infection-related revision and give direction to future complementation of the LROI with re-interventions due to PJI.

Study population: All patients who had primary THA or TKA in the included institutions will be followed up for 12 months until the end of the observation period (June 2027) or until the date of revision for infection, revisions for other indication, death or end of follow-up.

Main study parameters/endpoints: Related to the study objectives, the main study endpoints are as follows:

1. The percentage of hospitals that adopt to the new guideline and the time these hospitals take to do so.
2. The relative amount of revisions surgeries due to infection reported in the LROI and retrieved with CTcue, compared in the periode one year before implementation of the new guideline and one year after implementation of the new guideline.
3. The cost per antibiotic dose and the costs related to the extended hospital admission, compared between single-dose and multi-dose perioperative antibiotic prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

- Patients undergoing primary Total Hip Arthroplasty or primary Total Knee Arthroplasty

Exclusion Criteria:

- Patients undergoing Revision Hip Arthroplasty or Revision Knee arhtroplasty

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients undergoing Total Hip Arthroplasty and Total Knee Arthroplasty
Sampling Method: Probability Sample
Enrollment: 70000 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
The percentage of hospitals that adopt to the new guideline and the time these hospitals take to do so. | 2 years
The relative amount of revisions surgeries due to infection reported in the LROI and retrieved with CTcue, compared in the periode one year before implementation of the new guideline and one year after implementation of the new guideline. | 2 years
The cost per antibiotic dose and the costs related to the extended hospital admission, compared between single-dose and multi-dose perioperative antibiotic prophylaxis. | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- OLVG Hospital, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No